CLINICAL TRIAL: NCT06022705
Title: Evaluation of the Effect of APFEL Risk Score and Fasting Periods on Postoperative Nausea and/or Vomiting
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Collaborators: Tarsus University (Other)
Responsible Party: Principal Investigator, Derya Gezer, Assistant Profesor, Tarsus University
Other Study IDs: TarsusU
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Nausea, Postoperative; Vomiting, Postoperative; APFEL RİSK SCORE
Keywords: APFEL Risk Score,; Postoperative Nausea and Vomiting; Preoperative Fasting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study, it is aimed to determine the effect of Apfel risk score and fasting times on postoperative nausea and vomiting (PONV).

DETAILED DESCRIPTION:
PONV are common causes of delayed discharge. PONV; nausea and/or vomiting in the first 24 hours after surgery. The incidence of PONV after elective surgeries varies between 30-80% depending on anesthesia, type of surgery, and risk factors of the patient. PONV is not only an uncomfortable complication for the patient but is associated with significant patient dissatisfaction. It also includes dehydration, electrolyte imbalance, acid-base imbalance, pulmonary aspiration, pneumothorax, hypoxia, esophageal rupture, increased intracranial pressure, wound problems, bleeding, delayed oral intake, prolonged hospitalization, fatigue, anxiety, unexpected hospital readmission, increased medical costs. Therefore, the prevention and management of nausea and/or vomiting in the perioperative period in surgical patients is very important.

In the preoperative period, patients' risk of nausea and/or vomiting should be evaluated with standard measurement tools. The most commonly used is the Apfel risk score, including four risk factors. These; female gender, history of PONV and/or motion sickness, non-smoking, and postoperative opioid use. In the presence of 0, 1, 2, 3, and 4 risk factors, the incidence of PONV is approximately 10%, 20%, 40%, 60%, and 80%, respectively. It has been observed that the use of risk scoring for PONV significantly reduces the rate of nausea and vomiting in the postoperative period. The risk of PONV varies depending on the patient, the type of anesthesia and the surgery. Female gender, young age, non-smoking, history of PONV or motion sickness are important risk factors for PONV. Type of anesthesia, duration of administration, use of volatile anesthetics and nitrous oxide, and use of opioids in the perioperative period are among other risk factors. It has been reported that PONV is seen more frequently after laparoscopic, bariatric, gynecological surgery, and cholecystectomy.

In order to prevent the development of nausea-vomiting and aspiration pneumonia during and after the operation, patients should be fasted for a certain period of time before the operation. Fasting periods in the preoperative period should not be long enough to cause adverse outcomes in patients. It has been reported in the literature that long preoperative fasting periods do not prevent some complications, but on the contrary increase them. Therefore, it is emphasized that it is unnecessary to starve patients for a long time in the preoperative period. In the study of Hausel et al., it was reported that patients who were fasted for 12-24 hours before surgery had more nausea and vomiting in the postoperative period than patients who were fasted for a short time and were given oral carbohydrate-containing fluids. According to the results of different studies conducted in this area, it has been reported that reducing the preoperative fasting period eliminates the patient's feeling of thirst before the operation, reduces nausea and vomiting, alleviates anxiety, increases patient comfort, accelerates recovery, and significantly shortens the length of hospital stay. It is stated that a short pre-operative fasting period reduces the loss of nitrogen in the urine and prevents loss of muscle strength, reduces the feeling of anxiety and thirst before the operation, and increases patient comfort by reducing nausea and vomiting in the early postoperative period. It has been reported that there are limited clinical studies to explain the relationship between perioperative fasting time and PONV in terms of the level of evidence. In this respect, it is important to determine the relationship between risk factors preoperative fasting times, and PONV.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* To have applied for elective surgery,
* Being hospitalized 6 hours before the operation,
* American Society of Anesthesiologists (ASA) score I-III
* Not having a vision-hearing problem
* Not having chronic pain,
* No alcohol and/or substance addiction,

Exclusion Criteria:

* Performing emergency surgical intervention,
* Need for intensive care after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study will be composed of patients who applied for elective surgery to Çukurova University Medical Faculty Balcalı Training and Research Hospital General Surgery Clinic and Tarsus State Hospital General Surgery Clinic between the dates of the study. The sample, on the other hand, will consist of a total of 250 patients who comply with the selection criteria, agree to participate in the study, and are determined by power analysis.
  The sample of the study was carried out using an unknown population model. The data obtained from the study of Weibel et al. (2020) were used for the effect size to be used in the calculation of the sample number (Weibel et al., 2020).
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Determining the risk of posoperative nausea and vomiting. | 24 hours
  APFEL risk score. It is a valid tool to assess PONV and/or motion sickness, non-smoking status, and postoperative opioid use. Accordingly, 0-1 indicates low, 2-3 moderate and ≥3 high risk for ASBK. Accordingly, 0-1 indicates low risk, 2-3 moderate and ≥3 high risk for ASBK. In the presence of 0, 1, 2, 3 and 4 risk factors, the incidence of ASBK was reported as 10%, 20%, 40%, 60% and 80%, respectively.
Determination of postoperative nausea and vomiting. | 24 hours
  Nausea and Vomiting Evaluation Form. In our study, ASBK status will be evaluated as "Yes/No" at 0, 2, 4, 8, 12 and 24 hours using the Nausea and Vomiting Evaluation Form.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Results regarding the relationship between APFEL risk score fasting times and PONV will be shared. However, personal information will not be shared.

REFERENCES:
- [Background] Apfel CC, Heidrich FM, Jukar-Rao S, Jalota L, Hornuss C, Whelan RP, Zhang K, Cakmakkaya OS. Evidence-based analysis of risk factors for postoperative nausea and vomiting. Br J Anaesth. 2012 Nov;109(5):742-53. doi: 10.1093/bja/aes276. Epub 2012 Oct 3. PMID 23035051
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Wan KM, Carter J, Philp S. Predictors of early discharge after open gynecological surgery in the setting of an enhanced recovery after surgery protocol. J Obstet Gynaecol Res. 2016 Oct;42(10):1369-1374. doi: 10.1111/jog.13045. Epub 2016 Jun 29. PMID 27353883
- [Background] Parrish RH 2nd, Findley R, Elias KM, Kramer B, Johnson EG, Gramlich L, Nelson GS. Pharmacotherapeutic prophylaxis and post-operative outcomes within an Enhanced Recovery After Surgery (ERAS(R)) program: A randomized retrospective cohort study. Ann Med Surg (Lond). 2021 Dec 14;73:103178. doi: 10.1016/j.amsu.2021.103178. eCollection 2022 Jan. PMID 35003725
- [Background] Elvir-Lazo OL, White PF, Yumul R, Cruz Eng H. Management strategies for the treatment and prevention of postoperative/postdischarge nausea and vomiting: an updated review. F1000Res. 2020 Aug 13;9:F1000 Faculty Rev-983. doi: 10.12688/f1000research.21832.1. eCollection 2020. PMID 32913634
- [Background] Obrink E, Jildenstal P, Oddby E, Jakobsson JG. Post-operative nausea and vomiting: update on predicting the probability and ways to minimize its occurrence, with focus on ambulatory surgery. Int J Surg. 2015 Mar;15:100-6. doi: 10.1016/j.ijsu.2015.01.024. Epub 2015 Jan 29. PMID 25638733
- [Background] Veiga-Gil L, Pueyo J, Lopez-Olaondo L. Postoperative nausea and vomiting: physiopathology, risk factors, prophylaxis and treatment. Rev Esp Anestesiol Reanim. 2017 Apr;64(4):223-232. doi: 10.1016/j.redar.2016.10.001. Epub 2016 Dec 29. English, Spanish. PMID 28041609
- [Background] Cao X, White PF, Ma H. An update on the management of postoperative nausea and vomiting. J Anesth. 2017 Aug;31(4):617-626. doi: 10.1007/s00540-017-2363-x. Epub 2017 Apr 28. PMID 28455599
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Gecit S, Ozbayir T. Evaluation of Preoperative Risk Assessment and Postoperative Nausea and Vomiting: Importance for Nurses. J Perianesth Nurs. 2020 Dec;35(6):625-629. doi: 10.1016/j.jopan.2020.04.006. Epub 2020 Aug 7. PMID 32778493
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] American Society of Anesthesiologists Committee. Practice guidelines for preoperative fasting and the use of pharmacologic agents to reduce the risk of pulmonary aspiration: application to healthy patients undergoing elective procedures: an updated report by the American Society of Anesthesiologists Committee on Standards and Practice Parameters. Anesthesiology. 2011 Mar;114(3):495-511. doi: 10.1097/ALN.0b013e3181fcbfd9. No abstract available. PMID 21307770
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale R, Waitzberg DL, Bischoff SC, Singer P. ESPEN guideline: Clinical nutrition in surgery. Clin Nutr. 2017 Jun;36(3):623-650. doi: 10.1016/j.clnu.2017.02.013. Epub 2017 Mar 7. PMID 28385477
- [Background] Weibel S, Rucker G, Eberhart LH, Pace NL, Hartl HM, Jordan OL, Mayer D, Riemer M, Schaefer MS, Raj D, Backhaus I, Helf A, Schlesinger T, Kienbaum P, Kranke P. Drugs for preventing postoperative nausea and vomiting in adults after general anaesthesia: a network meta-analysis. Cochrane Database Syst Rev. 2020 Oct 19;10(10):CD012859. doi: 10.1002/14651858.CD012859.pub2. PMID 33075160
- See also: Preventable surgical harm in gynecologic oncology: optimizing quality and patient safety. — https://link.springer.com/content/pdf/10.1007/s13669-017-0226-y.pdf
- See also: REVIEW OF STUDIES EVALUATING THE EFFECT OF AROMATHERAPY ON THE MANAGEMENT OF POSTOPERATIVE NAUSEA AND VOMITING — https://dergipark.org.tr/tr/download/article-file/1528058
- See also: POSTOPERATIVE NAUSEA AND VOMITING — https://pdf.trdizin.gov.tr/pdf/SDVURXVWd0FQQnZodWYzK0VaSDk4SXlIMVFoZ3NJd1J3bUwvOGhjbGFrSDdXTEU3VkllWW9FNlpNNzk3UGpaV3FEMnAwaHJZa2UreG92eHNqbVA5U3dxZFRxcGdlbW0yMlkzemMxQndkS3VxejRKZE5HNVBTdkJObGFTckNROTZUZk4zYzBUUTh4b3ZOSjB0MmVHK2pVdFNkc0srRHpGck1xSU1mSFFMSnhZMmhzZnFIM3lUOVE5cUNudlhjcmN0eGNYOUQ1YWpIOW5wNW5KeG9GNytVdHJ3Sm5vUGU3RU1BajFoOHQ1amM2aUh1VGFvN0hRdjNjYUd1RTQ4UVFjWEFxeVM3VDBZMDJ3MUJBPT0
- See also: TSAR — https://www.tard.org.tr/assets/kilavuz/preoperatifdegerlendirme.pdf